CLINICAL TRIAL: NCT01971138
Title: Review of Surgical Site Infection Registration Routine at Surgery Departments in Sweden and Validation of One of the Used Routines
Status: Completed | Type: Observational
Sponsor: Halmstad County Hospital (Other)
Responsible Party: Principal Investigator, Claes Hjalmarsson, MD, PhD, Halmstad County Hospital
Other Study IDs: 121020-V02
Record Dates: First submitted 2013-08-28; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Surgical Site Infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical site infection registration: Is there a routine for SSI registration
  Interventions: Other: this is a survey

INTERVENTIONS:
Other: this is a survey

SUMMARY:
This study explores the routines of registration of surgical site infections (SSI) at different surgical centers in Sweden. It explores the sensitivity and specificity of the registration routines of SSI are at Halmstad County Hospital, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Clinics in Sweden that report tho the Swedish national register for Colorectal Cancer.

Exclusion Criteria:

* Clinics that dosen´t report.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgical clinics in Sweden.
Sampling Method: Non-Probability Sample
Dates: Start 2013-03; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
In which proportion do surgical clinics in Sweden register Surgical Site Infections | spring 2013
  A questionnaire will be sent to every surgical clinic in Sweden. This study will then summarize in what way the surgical clinics in Sweden perform their SSI surveillance.
In which proportion does the routine SSI registration at Halmstad County Hospital register the actual number of SSI´s. | up to four years
  Aiming to validate the SSI surveillance at Halmstad County Hospital. Patients who underwent elective colorectal resection between 2007-2008 were identified for inclusion in the study. A total of 66 patient were included. They were followed prospectively for four weeks and were controlled daily regarded SSI as a part of the study. After these four weeks the patients also filled a form regarding SSI. This group where then used as a control group. The results from the SSI registration routine at Halmstad County Hospital were then compared with the control group regarded SSI.

SECONDARY OUTCOMES:
Which method is used for routine registration of SSI´s in Sweden. | spring 2013
  A questionnaire will be sent to every surgical clinic in Sweden. This study will then summarize in what way the surgical clinics in Sweden perform their SSI surveillance.
How is the SSI classified in different hospitals in Sweden. | spring 2013
  A questionnaire will be sent to every surgical clinic in Sweden. This study will then summarize in what way the surgical clinics in Sweden perform their SSI surveillance.
How is the variation of SSI at the surgical clinic in Halmstad County Hospital, Sweden, the last 10 years. | for 10 years
  The study aims to do a statistical Analysis of the SSI surveillance material collected at the Halmstad County Hospital between 2002-2012. We want to know how big the variation is between years regarding SSI and if the statistics i good enough to draw conclusions from.
How large the difference have to be between in registered SSI frequency to surely detect a deviation in SSI presence | for 10 years
  The study aims to do a statistical Analysis of the SSI surveillance material collected at the Halmstad County Hospital between 2002-2012. We want to know how big the variation is between years regarding SSI and if the statistics i good enough to draw conclusions from.

CONTACTS AND LOCATIONS:
Overall Officials: Claes Hjalmarsson, MD, PhD, Principal Investigator — Halmstad County Hospital, Halmstad, Sweden
Locations (1):
- Halmstad County Hospital, Halmstad, Halland County, Sweden

REFERENCES:
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Smyth ET, Emmerson AM. Surgical site infection surveillance. J Hosp Infect. 2000 Jul;45(3):173-84. doi: 10.1053/jhin.2000.0736. PMID 10896795
- [Background] Degrate L, Garancini M, Misani M, Poli S, Nobili C, Romano F, Giordano L, Motta V, Uggeri F. Right colon, left colon, and rectal surgeries are not similar for surgical site infection development. Analysis of 277 elective and urgent colorectal resections. Int J Colorectal Dis. 2011 Jan;26(1):61-9. doi: 10.1007/s00384-010-1057-8. Epub 2010 Oct 5. PMID 20922541
- [Background] Malone DL, Genuit T, Tracy JK, Gannon C, Napolitano LM. Surgical site infections: reanalysis of risk factors. J Surg Res. 2002 Mar;103(1):89-95. doi: 10.1006/jsre.2001.6343. PMID 11855922
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Am J Infect Control. 1992 Oct;20(5):271-4. doi: 10.1016/s0196-6553(05)80201-9. No abstract available. PMID 1332552